CLINICAL TRIAL: NCT02273778
Title: A Pilot Study Investigating the Use of Co-registered 18FDG-PET-CT and MRI for Radiotherapy Planning in Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: MRI and PET-CT for Radiotherapy Planning for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CO10/9645; 11/YH/0212 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-10-14; First posted 2014-10-24 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Routine radiotherapy treatment plus MRI scan and PET-CT scan (Other)
  Interventions: Procedure: MRI Scan; Procedure: PET-CT Scan
- Routine radiotherapy treatment (Other)
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: MRI Scan
  Arms: Routine radiotherapy treatment plus MRI scan and PET-CT scan
Procedure: PET-CT Scan
  Arms: Routine radiotherapy treatment plus MRI scan and PET-CT scan
Other: No intervention
  Arms: Routine radiotherapy treatment

SUMMARY:
Radiotherapy is commonly used to treat advanced cancers of the head and neck, aiming for cure while preserving patients' quality of life including their ability to speak and swallow. In order to reduce the potentially major side effects of treatment, it is essential that the highest doses of radiotherapy are targeted to the main bulk of the tumour. At present a computerized tomography (CT) scan is used by the cancer specialist to identify the tumour for planning the radiotherapy treatment. The investigators know that other types of scan including magnetic resonance imaging (MRI) and positron emission tomography (PET) scans are better than CT scans at showing areas involved by the cancer. However, radiotherapy cannot be directly planned on these types of scans. The aim of this study is to explore whether PET and MRI scans can be combined with CT scans to more accurately identify the tumour target. In addition, this study will explore whether PETCT and MRI scans may used to adjust radiotherapy to how well a tumour is responding during a course of radiotherapy. If the radiotherapy planning process can be improved in these ways, the investigators hope future patients will benefit by more chance of cure with a reduction in the side effects of treatment. The study aims to recruit 16 patients. All patients within the study will undergo a PETCT and an MRI scan prior to starting treatment as part of the study. A subgroup of 8 patients will undergo additional imaging at two timepoints during the course of their radiotherapy. The study is noninterventional and patients' standard treatment will not be affected by their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* WHO Performance status 02
* Histologically proven squamous cell carcinoma of the head and neck region
* Clinical decision made to proceed with a course of radiotherapy of curative intent of 6670Gy in 3335 fractions over six and a half to seven weeks with or without concurrent chemotherapy
* Measurable primary tumour and/or locoregional metastatic lymph nodes on preradiotherapy imaging
* Able to provide fully informed written consent
* Able to lie flat for 1 hour
* Not be pregnant or breast feeding. Female patients of childbearing potential must agree to use effective contraception, be surgically sterile, or be postmenopausal.

Exclusion Criteria:

* Hypersensitivity to fluorine-18 FDG
* Hypersensitivity to iodinated contrast media or Gadolinium
* Poorly controlled diabetes
* Acute renal failure or moderate renal impairment (estimated glomerularb filtration rate < 30 mL/min)
* Contraindication to MRI imaging, including cardiac pacemaker or presence of MRI incompatible metalwork
* Claustrophobia precluding MRI imaging
* Uncontrolled pain
* Urinary incontinence
* Female patients must not be pregnant and if of child bearing age using adequate contraception
* Breast feeding
* Serious psychiatric comorbidity

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of utilising MRI images in head and neck radiotherapy planning. | 40-60 minutes
  Determine whether MRI images in head and neck radiotherapy can be used to modify the tumour target volume during radiotherapy.
Feasibility of utilising PET-CT images in head and neck radiotherapy planning. | 2 hours
  Determine whether PET-CT images in head and neck radiotherapy can be used to modify the tumour target volume during radiotherapy.